CLINICAL TRIAL: NCT04014582
Title: Communal Coping Intervention for Couples With Type 2 Diabetes
Brief Title: Taking Action: a Care for Type 2 Diabetes Intervention for Couples
Acronym: TACTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Melissa Zajdel, PhD Candidate Psychology, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY2019_00000227
Record Dates: First submitted 2019-06-26; First posted 2019-07-10 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes
Keywords: communal coping; couples coping; adjustment
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two groups, either the intervention or the control (diabetes education) condition
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly assigned to condition, and they will not be aware if they are in the intervention or control group. The control group is more than usual care, so they may also believe they are in the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communal Coping Intervention (Experimental): This group will participate in diabetes education + a communal coping based intervention.
  Interventions: Behavioral: Communal Coping Intervention
- Control (Active Comparator): This group will participate in diabetes education and an individual intervention.
  Interventions: Behavioral: Diabetes Education

INTERVENTIONS:
Behavioral: Communal Coping Intervention — This intervention aims to foster a shared appraisal and collaboration through: the discussion of past joint coping, education about communal coping (e.g. what it is and why it is beneficial), and discussions to foster the perception of diabetes as shared. Participants in the intervention group will also create collaborative action plans to increase collaboration. Couples in the intervention group will also receive two daily text messages-one a general reminder to engage in communal coping and the other one of the collaborative intentions they created during the in-person session. These couples will also receive a brief diabetes education.
  Arms: Communal Coping Intervention
Behavioral: Diabetes Education — Couples in the diabetes education group will receive a brief diabetes education and complete individual implementation intentions. Patients will create implementation intentions related to diabetes and partners will create implementation intentions that are not related to health.
  Other Names: Control
  Arms: Control

SUMMARY:
Communal coping consists of the appraisal of a problem as shared and collaboration to manage the problem. Among individuals with type 2 diabetes, self-report, daily diary, and observational measures of communal coping have been linked to better relationship and health outcomes. While communal coping has been linked to positive adjustment outcomes, there are no interventions that incorporate both components of communal coping theory; interventions often focus on collaborative strategies but do not emphasize a shared appraisal. However, focusing on the shared appraisal component of communal coping may be the critical component to affect change. The primary goal of this study will be to design an intervention that fosters both a shared appraisal and collaboration in individuals with type 2 diabetes. The second goal is to explore two potential mechanisms that may drive the links of the intervention to outcomes-perceived emotional responsiveness and self-efficacy.

DETAILED DESCRIPTION:
Participants will be 60 couples recruited from a previous research study in which one person has type 2 diabetes. We will recruit 60 couples based on power analyses of collaboration based interventions. The design will be a two-group pretest-posttest design in which couples will be randomly assigned to one of two conditions: communal coping or diabetes education. All couples will engage in 1) an in-person session, 2) a 7-day daily diary protocol, and 3) a phone call follow-up 1 month later. All participants will come into the laboratory at Carnegie Mellon University to complete a baseline questionnaire and listen to a brief diabetes education from the American Association of Diabetes Educators. Couples in the intervention group will then participate in the communal coping intervention. This intervention aims to foster a shared appraisal and collaboration through: the discussion of past joint coping, education about communal coping (e.g. what it is and why it is beneficial), and discussions to foster the perception of diabetes as shared. Participants in the intervention group will also create collaborative action plans to increase collaboration-collaborative intentions have been shown to successfully impact health outcomes for patients with type 2 diabetes. Couples in the intervention group will also receive two daily text messages-one a general reminder to engage in communal coping and the other one of the collaborative intentions they created during the in-person session.

There will be two follow-up periods after this in-person session. First, all couples will answer daily questionnaires over a 7-day period starting the day after the in-person session. The second follow-up will be one month after the daily diary period, when couples will receive a follow up phone call to assess how the primary outcomes of interest changed over a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

* One person must have type 2 diabetes.
* Must be married or cohabitating for at least 1 year with a partner
* Must have access to internet to participate (required for daily diary component).

Exclusion Criteria:

* Both persons cannot have type 2 diabetes
* Must not have any other major comorbidities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | Depressive symptoms will be measured at baseline and 1 month after the intervention.
  Depressive symptoms will be measured via the 10 item CESD scale which range from 1 none of the time to 4 most of the time. This self-report questionnaire will be assessed for both patient and spouse. Higher numbers represent more depressive symptoms.
Change in life satisfaction | Life satisfaction will be measured at baseline and 1 month after the intervention.
  Life satisfaction will be measured via the Satisfaction with Life scale which range from 1 strongly disagree to 7 strongly agree. Higher numbers represent more life satisfaction. Both patients and spouses will report on life satisfaction.
Change in perceived stress | Perceived stress will be measured at baseline and 1 month after the intervention.
  Perceived stress will be measured via the 4 item Perceived Stress Scale which ranges from 1 never to 5 very often. Both patients and spouses will complete this self-report questionnaire.
Change in relationship satisfaction--QMI | Relationship satisfaction--QMI will be measured at baseline and 1 month after the intervention.
  Relationship satisfaction will be measured via the Quality of Marriage Index. This self-report scale ranges from 1 strongly disagree to 7 strongly agree. Both patients and spouses will complete this self-report questionnaire.
Change in relationship satisfaction--PAIR | Relationship satisfaction will be measured at baseline and 1 month after the intervention.
  Relationship satisfaction will also be measured via the Personal Assessment of Intimacy in Relationships scale. This scale will be assessed from 1 strongly disagree to 7 strongly agree. Both patients and spouses will complete this questionnaire.
Change in diabetes self-care | Diabetes self-care will be measured at baseline and 1 month after the intervention.
  Diabetes self-care will be measured via the summary of diabetes self care activities. Patients will report on their own self care and spouses will report on their perceptions of the patient's self-care. The items in the SDSCA have varying scales based on the question, but higher numbers reflect greater self-care.

SECONDARY OUTCOMES:
Change in perceived emotional responsiveness | Perceived emotional responsiveness will be measured at measured at baseline and 1 month after the intervention.
  Perceived emotional responsiveness measures the extent to which a spouse feels appropriately supported and understood by the partner. The items used in this scale are modified versions used by Fekete et al. 2007. The scale ranges from 1 not at all to 4 very much. Negative items will be reversed scored so the total scale reflects greater perceived emotional responsiveness for both patients and spouses.
Change in generalized self-efficacy | Self-efficacy will be measured at baseline and 1 month after the intervention.
  Self-efficacy will be measured via the new generalized self-efficacy scale. This scale ranges from 1 strongly disagree to 5 strongly agree. Higher numbers reflect greater self-efficacy. Both patients and spouses will report generalized self efficacy.
Change in diabetes specific self-efficacy | Self-efficacy will be measured at baseline and 1 month after the intervention.
  Self-efficacy will be measured via the diabetes specific self-efficacy scale. Patients will report their confidence in their abilities to take care of certain diabetes related behaviors. Spouses will report on their confidence of the patient's ability to engage in diabetes self care behaviors. The scale ranges from 0-100.

OTHER OUTCOMES:
Daily mood | Daily mood will be measured over a 7 day daily diary period.
  Daily mood will be assessed via a modified version of the PANAS scale. These items will be assessed via 1 not at all to 5 a lot. Negative items will be reversed coded so that greater overall scale scores reflect more positive daily mood. Both patients and spouses will report on daily mood.
Daily self-care behaviors. | Daily mood will be measured over a 7 day daily diary period.
  Daily mood will be assessed via a modified version of SDSCA scale. The response scale for these items will vary based on the question. Higher scores will reflect more daily self-care behaviors. Patients will report on their own self-care behaviors and spouses will report on the patient's self-care behavior.
Daily relationship satisfaction | Daily relationship satisfaction will be measured over a 7 day daily diary period.
  Daily relationship satisfaction will be assessed via a shortened and modified version of the QMI scale. Numbers range from 1-7 with higher numbers reflect greater relationship satisfaction. Both patients and spouses will report on relationship satisfaction.
Daily diabetes self-efficacy | Daily diabetes self efficacy will be measured over a 7 day daily diary period.
  Daily diabetes self-efficacy will be assessed via shortened and modified versions of diabetes self-efficacy scale. Scale ranges from 0-100 with higher numbers representing more self-efficacy. Patients will report how confident they felt that day regarding their diabetes management that day.
Daily self-efficacy | Daily self efficacy will be measured over a 7 day daily diary period.
  Daily self-efficacy will be assessed via shortened and modified versions of the new generalized self-efficacy scale. Higher numbers will reflect greater self-efficacy. Both patients and spouses will report on daily generalized self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Carnegie Mellon Universityl, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared on CMU's KiltHub website. Built upon the figshare platform, KiltHub collects, preserves, and provides stable, long-term global open access to a wide range of research data and scholarly outputs. All datasets and scholarly outputs published on KiltHub receive their own DOI, recommended citation, a machine-readable copyright license, and is indexed in Google. Cleaned data, codebook, and documents that explain the file naming schema and files available will be published on KiltHub.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The above data and materials will be made available upon first publication from the study.
Access Criteria: The data will openly accessible and discoverable with a unique DOI on CMU's Kilthub data sharing platform.